CLINICAL TRIAL: NCT01101685
Title: Blood Oxygen Level Dependent (BOLD) Responses During Emotional and Cognitive Processing in Dysphoric and Non-dysphoric Participants and Their Modulation by a Pharmacological Probe of Serotonin Function
Brief Title: Neural Responses and Dysphoria: Modulation by a Pharmacological Probe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: P1vital Limited (Industry); University of Manchester (Other); Institute of Psychiatry, London (Other)
Responsible Party: Professor Guy Goodwin, Oxford University, Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: P1V-DEP-CT02-09
Record Dates: First submitted 2010-03-31; First posted 2010-04-12 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Dysphoria
Keywords: non-dysphoric; Dysphoric
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram (Active Comparator): 7 days dosing at 10mg per day
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): 7 days dosing at 10mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 7 days dosing of 10mg per day
  Arms: Escitalopram
Drug: Placebo — 7 days dosing at 10mg daily
  Arms: Placebo

SUMMARY:
This study aims to improve understanding of how people with low mood and negative feelings (known as dysphoric) may be different from people with normal mood and feelings (nondysphoric) when responding to a variety of social and emotional information. The study will look at the patterns of activity in peoples' brains in situations (presented as a battery of tests) after treatment with a medicine (escitalopram) or a placebo. The results from this study will help to gather information about the effectiveness of the various tests being used in this study in detecting any changes due to treatment with an antidepressant. Half the volunteers taking part in this study will be dysphoric (mildly depressed) whilst the other half of volunteers will be healthy volunteers. It is hoped that the results of this study will provide guidance for assessing effectiveness of new medicines and potentially help with the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 45 years, inclusive at Randomisation visit.
* Fluent English speakers.
* Beck Depression Inventory (BDI) score of 05 or ≥10 at both Screening and Randomisation visits.
* Hamilton Depression Rating Scale (HAMD)score of <24 at both Screening and Randomisation visits.
* Healthy at Screening visit as determined by a physician.
* Female participants should be surgically sterile or abstinent or, if sexually active, be practising an effective method of birth control.
* Acceptable weight as defined by body mass index (BMI) range of 18 to 30 kg/m², inclusive.
* Normotensive with sitting (5 minutes) blood pressure between the range of 100 to 140 mmHg systolic, inclusive and 60 to 90 mmHg diastolic, inclusive at Screening.
* Non smoker or light smoker (≤ 5 cigarettes per day).
* Participants must have signed the Informed Consent Form.
* Participants providing a genetic sample must have signed the DNA consent.

Exclusion Criteria:

* History of alcohol or substance dependence within the last 6 months.
* Consumption of large amounts of caffeinated drinks.
* Relevant history or presence upon clinical examination, of cardiac, ophthalmologic, pulmonary, endocrine (diabetes),cancer, blood disease, gastrointestinal, hepatic or renal disease or other condition.
* History or presence of significant neurological or psychiatric conditions. Exceptions to this are participants with a history of depression for the dysphoric group. Participants with generalised anxiety disorder or other anxiety disorders may be entered at the discretion of the Investigator.
* Participants who, in the opinion of the Investigator, are at risk of suicide.
* Any use of sedative hypnotics, including benzodiazepines, zolpidem or zopiclone within the last 3 months prior to Randomisation visit.
* Any use of medications for depression in the last three months prior to Randomisation visit.
* Have received prescribed medication within 14 days prior to Randomisation visit (apart from the contraceptive pill).
* Have received over-the-counter (OTC) medicine within 48 hours prior to Randomisation visit.
* Have received an experimental drug and/or used an experimental medical device within 30 days of Randomisation visit or within a period less than 5 times the drug's half life, whichever is longer.
* If female: are pregnant or are trying to get pregnant or are currently breast feeding.
* History of, or current condition of, migraine headaches or have undergone operations to the head.
* Significant hearing impairment.
* Significant visual impairment or history of ocular treatment.
* Lefthanded.
* Previous experience of the emotional test battery experimental procedures.
* Unable to comply with magnetic resonance (MR) Patient Declaration.
* Involvement in an emergency (medically emergent) situation between Screening and Randomisation visits.
* Surgery between Screening and Randomisation visits.
* Unable or unwilling to comply with study procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) responses during emotional and cognitive processing | 1 day

SECONDARY OUTCOMES:
Validating the sensitivity of dysphoric verses nondysphoric reactions to cognitive and emotional stimuli in detecting antidepressant drug effects. | 1 day
  Using tests of cognitive and emotional processing, specially:
  Emotional Counting Stroop Emotional Encoding Task Sad Music Visual checkerboard Facial Expression Processing Dot-Probe N-Back digit Symbol substitution California Verbal Learning Test Depression Realism Task
Genetic influences on the processing of cognitive and emotional stimuli. | 6 months to 1 year after study completion
Relationship between BOLD fMRI signals and emotional processing using a biomarker test battery | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Guy Goodwin, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, Oxford, United Kingdom